CLINICAL TRIAL: NCT02015572
Title: Retention in Physically Demanding Jobs With Low Back Pain: A Randomised Controlled Trial (GoBack)
Acronym: GoBack
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Frederiksberg University Hospital (Other)
Collaborators: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Bjarke Brandt Hansen, MD, Frederiksberg University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GoBack-001
Record Dates: First submitted 2013-11-29; First posted 2013-12-19 (Estimated); Last update posted 2017-02-13 (Actual); Status verified 2017-02

CONDITIONS: Low Back Pain
Keywords: Low back pain; Return to work; Sickness absence; Rehabilitation; Occupational intervention
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Occupational intervention (Experimental): Early coordinated occupational intervention. Supervision in physically activities by a physiotherapist.
  Interventions: Behavioral: Occupational intervention
- Usual care (Active Comparator): Intervention from the patient's general physician.
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: Occupational intervention — Early coordinated occupational intervention and supervision in physically activities by a physiotherapist.
  Arms: Occupational intervention
Other: Usual care — Intervention from physiotherapist, chiropractor, rheumatologist coordinated by the patient's general physician
  Arms: Usual care

SUMMARY:
Low back pain (LBP) is a recognized public health problem with high life time prevalence. Medical treatment may reduce the physical and mental discomfort, while it has not been able to improve the possibilities for retaining or return patients with LBP to work.

This is an occupational intervention study for patients with LBP and physically demanding work, who are at risk of drop out of labour; a randomized controlled trial designed to test the effectiveness of an early intervention for retaining subjects with LBP attached to the labour marked. A work place modification intervention combined with moderate physical activity is given in the intervention group additional to LBP treatments according to best practice recommendations for general practice.

The study population consists of patients in self-reported physically demanding, who are sick listed or at risk of sick leave due to LBP. Outcome will continually be collected during the intervention as well as 6 and additionally at 12 months follow up.

The primary aim is to evaluate if an occupational intervention with focus on early workplace orientated counselling and work place intervention can retain subjects with physically demanding work and LBP in gainful employment to prevent/reduce the sick leave due to LBP.

The secondary aims are to identify prognostic factors of an occupational intervention using the baseline and follow-up participant-rated outcomes: pain, physically function, generic health status, fear avoidance behaviours, job satisfaction, work-ability, satisfaction with intervention, clinical examination and MRI findings. Among these variables, we also aim to identify subjects, who will benefit from such an occupational intervention, and the subjects, who already have a good prognosis and therefore have no need for a larger scale intervention.

DETAILED DESCRIPTION:
Eligible participants are: 1) 18-65 years of age; 2) current episode of 2-4 weeks of LBP; 3) self-reported physically demanding work; 4) express concerns about the ability to maintain their current job.

The exclusion criteria are: 1) pregnancy; 2) server somatic or psychiatric diseases; 3) cancer or metastatic disease

ELIGIBILITY:
Inclusion Criteria:

* Working age adults 18-65
* Low back pain (current episode of 2-4 weeks)
* Self-reported physically demanding work
* Sick-listed or at risk
* Speak, read and understand Danish
* Accept workplace visit by the occupational physicians
* Be in gainful employment for at last 30 hours/week

Exclusion Criteria:

* Severe somatic or psychiatric comorbidity
* Pregnancy
* Cancer or metastatic disease
* LBP treatment or referral to outside providers (e.g. back-surgery)
* Contraindications for having a MRI.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2016-01; Primary Completion 2016-06 (Actual); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Accumulated duration of self-assessed sick leave due to LBP | 6 months

SECONDARY OUTCOMES:
Changes in pain level | 6 months
  Pain will be evaluated by using the 13 items Pain-Detect questionnaire, which includes measurements of LBP on an ordinal, 11-point numerical rating scale (NRS: 0 = no LBP; 10 = worst LBP possible).
Changes in Fear Avoidance Beliefs scores | 6 months
  Both Fear Avoidance Beliefs Work Subscale and Physical Activity subscale (questionnaires) will be measured.
Change in Disability | 6 months
  The 24-item Roland Morris Disability Questionnaire will measure participant-rated LBP disability.
Satisfaction with the intervention | 6 months
  Measured on an 11-point NRS with the anchors "not at all satisfied" to "extremely satisfied".

OTHER OUTCOMES:
Accumulated duration of self-assessed sick leave due to LBP | 12 months
MRI findings | Baseline
  Degree of degenerative MRI findings in the lumbar spine predicts outcome (sick leave)
Predictors of outcome | Baseline
  Baseline questionnaires scores (Pain categorization (PainDETECT®), Numeric Pain Rating Scale (NPRS), Fear Avoidance Beliefs, 36-item short-form health-survey (SF36) and Roland Morris Disability) are associated with outcome (sick leave).

CONTACTS AND LOCATIONS:
Overall Officials: Ann Kryger, MD, PhD, Principal Investigator — University Hospital Frederiksberg and Bispebjerg
Locations (1):
- The Parker Institute, Department of Rheumatology, Copenhagen University Hospital, Bispebjerg and Frederiksberg Hospital, Copenhagen, Frederiksberg, Denmark

REFERENCES:
- [Background] Jensen C, Jensen OK, Nielsen CV. Sustainability of return to work in sick-listed employees with low-back pain. Two-year follow-up in a randomized clinical trial comparing multidisciplinary and brief intervention. BMC Musculoskelet Disord. 2012 Aug 25;13:156. doi: 10.1186/1471-2474-13-156. PMID 22920158
- [Derived] Rosenberg NR, Petersen SB, Begtrup LM, Flachs EM, Petersen JA, Hansen BB, Kirkeskov L, Bliddal H, Christensen R, Kristensen LE, Fournier GL, Kryger AI. Early Occupational Intervention for People with Low Back Pain in Physically Demanding Jobs: 1-year Follow-up Results of the Randomized Controlled GOBACK Trial. Spine (Phila Pa 1976). 2021 Mar 15;46(6):347-355. doi: 10.1097/BRS.0000000000003793. PMID 33181779
- [Derived] Hansen BB, Kirkeskov L, Begtrup LM, Boesen M, Bliddal H, Christensen R, Andreasen DL, Kristensen LE, Flachs EM, Kryger AI. Early occupational intervention for people with low back pain in physically demanding jobs: A randomized clinical trial. PLoS Med. 2019 Aug 16;16(8):e1002898. doi: 10.1371/journal.pmed.1002898. eCollection 2019 Aug. PMID 31419219
- [Derived] Petersen J, Kirkeskov L, Hansen BB, Begtrup LM, Flachs EM, Boesen M, Hansen P, Bliddal H, Kryger AI. Physical demand at work and sick leave due to low back pain: a cross-sectional study. BMJ Open. 2019 May 22;9(5):e026917. doi: 10.1136/bmjopen-2018-026917. PMID 31122982
- [Derived] Hansen BB, Kirkeskov L, Christensen R, Begtrup LM, Pedersen EB, Teilya JF, Boesen M, Fournier GL, Bliddal H, Kryger AI. Retention in physically demanding jobs of individuals with low back pain: study protocol for a randomised controlled trial. Trials. 2015 Apr 16;16:166. doi: 10.1186/s13063-015-0684-3. PMID 25887302
- See also: Department of Occupational and Environmental Medicine, Copenhagen University, Hospital Bispebjerg and Frederiksberg — http://www.bispebjerghospital.dk/menu/Afdelinger/Kliniske+afdelinger/Arbejds+og+Miljoemedicinsk+Afdeling/?siu=true
- See also: The Parker Institute, Department of Rheumatology, Copenhagen University Hospital, Bispebjerg and Frederiksberg Hospital — http://www.parkerinst.dk/